CLINICAL TRIAL: NCT06625684
Title: Key Longitudinal Associations With Risk and Glioblastoma Outcomes
Acronym: Key LARGO
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Glioblastoma Research Organization (Unknown); StacheStrong (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00114859
Record Dates: First submitted 2024-09-25; First posted 2024-10-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; genetic predisposition to disease; risk factors; quality of life; questionnaires; blood sample; adult brain cancer; observational study; personal medical history; survival outcomes; cancer epidemiology; genetics, medical; immunologic factors; patient outcomes; health history; occupational exposure
MeSH Terms: conditions — Glioblastoma; Genetic Predisposition to Disease; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will retain peripheral blood samples collected from participants. These samples will be used for extracting DNA to analyze genetic factors related to glioblastoma. Additionally, any remaining biological material from these blood samples may be used for other relevant analyses as needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Glioblastoma: This group consists of adults diagnosed with glioblastoma, a type of aggressive brain tumor. Participants are observed to identify factors influencing their outcomes, including genetic, immunologic, and personal medical history factors. The study aims to explore how these factors impact survival rates and quality of life in this patient population. There are no specific interventions. Instead, the focus is on analyzing survey data and biological samples to understand risk factors and disease progression.

SUMMARY:
The goal of this observational study is to find out what factors affect the health and risks in adults with glioblastoma (GBM), a grade 4 brain cancer.

The main questions it aims to answer are:

* How do genetic and immune system factors impact survival and quality of life in GBM patients?
* What occupational and medical history factors are linked to the risk of getting GBM?

Participants will:

* Fill out an online survey about their medical history and lifestyle.

Participants will have the chance to give a blood sample (from the outer arm) for genetic and immune system testing. Blood samples will be given using a home collection kit provided by the study team.

DETAILED DESCRIPTION:
This observational study aims to investigate the various factors influencing outcomes and risks in adults diagnosed with glioblastoma (GBM). Glioblastoma is a highly aggressive and malignant brain tumor, and understanding the factors that affect patient outcomes is crucial for improving management strategies and patient care.

The study employs a case-only design where participants will be followed over time to observe how different factors affect their health outcomes. Participants will be selected based on their diagnosis of glioblastoma and will be included in the study regardless of current treatment status or disease stage.

Findings from this study are expected to provide valuable insights into the factors affecting glioblastoma outcomes and may contribute to the development of personalized treatment strategies and risk assessment tools for better management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Pathologically-confirmed diagnosis of glioblastoma multiforme (GBM) or grade 4 brain tumor
* Participant is accessible for follow-up (has a working email address)
* Participant is willing and able to comply with the study requirements

Exclusion Criteria:

* Those who cannot read either English or Spanish
* Those who cannot view an online survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit glioblastoma (GBM) patients from the general population through social media and email listservs. Recruitment efforts will be supported by GBMRO, StacheStrong, and the Duke Preston Robert Tisch Brain Tumor Center. These organizations will disseminate study information via electronic communications to their GBM patient listservs and promote the study on social media platforms such as Facebook and Twitter. The study aims to enroll a diverse population of GBM patients from around the world, ensuring broad representation across various demographics and regions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-12-10 (Estimated); Study Completion 2029-12-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of enrollment until date of death from any cause as submitted by caregiver, up to 60 months
  Overall survival will be estimated using patient-reported date of diagnosis and assessed in three month intervals until patients are reported as deceased or are lost to follow-up
Functional Well-being as measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire | At time of study enrollment
  Estimated using the functional well-being subscale of the FACT-Br questionnaire. The score ranges from 0 to 28, where a higher score indicates greater functional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Quinn Ostrom, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No